CLINICAL TRIAL: NCT00698516
Title: An Open-label, Multicenter, Non-comparative, Phase II Study of Oral Topotecan in Combination With Bevacizumab for Second-line Treatment in Subjects With Relapsed Small-cell Lung Cancer (SCLC)
Brief Title: Study of Oral Topotecan With Bevacizumab for Recurrent Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104864/111127
Record Dates: First submitted 2008-06-16; First posted 2008-06-17 (Estimated); Results first posted 2011-02-03 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2011-03

CONDITIONS: Recurrent Small-cell Lung Cancer (SCLC); Lung Cancer, Small Cell
Keywords: Bevacizumab; Small Cell Lung Cancer (SCLC); Topotecan
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan; Capsules; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label, Single arm (Experimental): Oral topotecan + IV Bevacizumab
  Interventions: Drug: Oral Hycamtin (topotecan) Capsules + IV Avastin (bevacizumab)

INTERVENTIONS:
Drug: Oral Hycamtin (topotecan) Capsules + IV Avastin (bevacizumab) — 2.3 mg/m2 daily x 5 oral topotecan and 15 mg/kg IV bevacizumab on day 1 of every 21 days cycle.

SUMMARY:
Combination of Hycamtin (topotecan) and Avastin (bevacizumab) could allow killing of both endothelial and neoplastic cells. We postulate that addition of bevacizumab to topotecan will increase delivery of topotecan to tumor cells and may enhance activity of topotecan in patients with previously treated small cell lung cancer and improve progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of SCLC.
* First recurrence of SCLC after therapy with one prior chemotherapy regimen at initial diagnosis.
* Relapsed SCLC of any duration (both sensitive and resistant relapse).
* ECOG performance status of </= 2.
* Adequate bone marrow reserve, hepatic, renal, and cardiovascular function.
* No prior therapy with bevacizumab or any other VEGF inhibitor or topotecan

Exclusion Criteria:

* Uncontrolled emesis, regardless of etiology.
* Active uncontrolled infection.
* GI conditions or drugs that could impact absorption of oral topotecan.
* Known hypersensitivity to any component of topotecan capsule or compounds chemically related to topotecan.
* Uncontrolled hypertension with BP>150/100.
* Prior h/o hypertensive crisis or encephalopathy.
* NYHA Grade II or greater congestive heart failure.
* H/O myocardial infarction within 6 months.
* H/O stroke or TIA within 6 months.
* H/O thrombotic or hemorrhagic disorders.
* Clinically significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days.
* Anticipation of need for major surgical procedure during the study.
* Minor surgical procedures within 7 days prior to treatment start (placement of vascular access devices is permitted).
* H/O abdominal fistula, GI perforation, or intra-abdominal abscess within prior 6 months. Serious, non-healing wound, active ulcer, or untreated bone fracture. - H/O hemoptysis within prior 1 month.
* Concurrent radiotherapy.
* H/O whole lung radiation within 90 days prior to start of treatment.
* Presence or h/o central nervous system or brain metastases.
* H/o another malignancy other than SCLC.
* Concurrent chemotherapy, immunotherapy, or investigational therapy for the treatment of small cell lung cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- United States (15):
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Naples, Florida
  - GSK Investigational Site, Athens, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Madison, Wisconsin

REFERENCES:
- [Derived] Spigel DR, Waterhouse DM, Lane S, Legenne P, Bhatt K. Efficacy and safety of oral topotecan and bevacizumab combination as second-line treatment for relapsed small-cell lung cancer: an open-label multicenter single-arm phase II study. Clin Lung Cancer. 2013 Jul;14(4):356-63. doi: 10.1016/j.cllc.2012.12.003. Epub 2013 Feb 4. PMID 23391616

RESULTS

PARTICIPANT FLOW:
Groups:
- Topotecan and Bevacizumab: Participants were to receive oral topotecan 2.3 milligrams (mg)/meters squared (m^2)/day for 5 consecutive days (Days 1 to 5) and intravenous (IV) bevacizumab 15 mg/kilograms (kg) on Day 1 of each 21-day cycle. Treatment was to be continued for up to 8 cycles (a minimum of 4 cycles was recommended) or until disease progression or development of unacceptable toxicity, whichever occurred first. Prior approval from GlaxoSmithKline's study physician was needed for participants who required treatment beyond 8 cycles.
Period: Overall Study
Arm/Group | Topotecan and Bevacizumab
Started | 50
Completed | 45
Not Completed | 5
Not completed — Study Termination | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Topotecan and Bevacizumab
Number analyzed (Participants) | 50
Age Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 24
Race/Ethnicity, Customized [Number; unit: participants]
  White | 43
  African American/African Heritage | 6
  White and Mixed Race | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-free Survival (PFS) at 3 Months
Description: PFS = time from initiation of drug to time of first disease progression/death due to any cause. Progression assessed using Response Evaluation Criteria (RECIST): >=20% increase in sum of longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since treatment started, or appearance of new lesion(s). If participant did not progress or die, the time of initiation of post-treatment anti-cancer therapy or time of last contact used. PFS at 3 months calculated by taking the Kaplan-Meier (KM) estimate at 90 days from the initiation of treatment. SE = standard error.
Time Frame: 3 months
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of study medication
Measure: Number; unit: percentageof participants
Arm/Group | Topotecan and Bevacizumab
Number analyzed (Participants) | 50
percentageof participants | 65
Statistical Analysis 1: Comparison: Topotecan and Bevacizumab; Test type: Superiority or Other; p = 0.017, Z statistic — Historical data in target population showed 3-month PFS rates of <=50%. Oral topotecan with IV bevacizumab would provide clinically meaningful improvement in 3-month PFS if it could demonstrate a 40% improvement relative to the historical data; Z statistic was used to reject the null hypothesis provided Z>=1.65, where Z = (KM estimate at 3 months - null hypothesis value [50%])/Greenwood SE; Greenwood variance = 65.0, 95% CI 2-sided [49.3 to 76.9], Standard Error of Mean 7.07

2. Secondary Outcome: PFS - Overall
Description: Progression-free survival at any site was defined as the time from initiation of investigational product to the time of first documented disease progression or death due to any cause. Progression was assessed using the RECIST guidelines: >= 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since treatment started, or appearance of new lesion (s). For participants who did not progress or die, the time of initiation of post-treatment anti-cancer therapy or the time of last contact was used.
Time Frame: Baseline to disease progression or death (up to 82.4 weeks)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Topotecan and Bevacizumab: Resistant Participants: Participants were to receive oral topotecan 2.3 milligrams (mg)/meters squared (m^2)/day for 5 consecutive days (Days 1 to 5) and intravenous (IV) bevacizumab 15 mg/kilograms (kg) on Day 1 of each 21-day cycle. Treatment was to be continued for up to 8 cycles (a minimum of 4 cycles was recommended) or until disease progression or development of unacceptable toxicity, whichever occurred first. Prior approval from GlaxoSmithKline's study physician was needed for participants who required treatment beyond 8 cycles. The time to progression from the end of prior chemotherapy was <= 90 days; therefore, these participants were termed "resistant".
- Topotecan and Bevacizumab: Sensitive Participants: Participants were to receive oral topotecan 2.3 milligrams (mg)/meters squared (m^2)/day for 5 consecutive days (Days 1 to 5) and intravenous (IV) bevacizumab 15 mg/kilograms (kg) on Day 1 of each 21-day cycle. Treatment was to be continued for up to 8 cycles (a minimum of 4 cycles was recommended) or until disease progression or development of unacceptable toxicity, whichever occurred first. Prior approval from GlaxoSmithKline's study physician was needed for participants who required treatment beyond 8 cycles. The time to progression from the end of prior chemotherapy was >90 days; therefore, these participants were termed "sensitive".
- Topotecan and Bevacizumab: All Participants: Participants were to receive oral topotecan 2.3 milligrams (mg)/meters squared (m^2)/day for 5 consecutive days (Days 1 to 5) and intravenous (IV) bevacizumab 15 mg/kilograms (kg) on Day 1 of each 21-day cycle. Treatment was to be continued for up to 8 cycles (a minimum of 4 cycles was recommended) or until disease progression or development of unacceptable toxicity, whichever occurred first. Prior approval from GlaxoSmithKline's study physician was needed for participants who required treatment beyond 8 cycles. This groups consists of both resistant and sensitive participants.
Arm/Group | Topotecan and Bevacizumab: Resistant Participants | Topotecan and Bevacizumab: Sensitive Participants | Topotecan and Bevacizumab: All Participants
Number analyzed (Participants) | 23 | 27 | 50
weeks | 12.64 [6.43 to 21.43] | 27.14 [16.14 to 32.57] | 17.43 [13.14 to 25.00]

3. Secondary Outcome: Number of Participants With Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD)
Description: Tumor response was determined using the RECIST guidelines.CR, disappearance of all target lesions; PR, >=30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; SD, neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since treatment started; PD, >=20% increase in sum of LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Baseline to disease progression or death (up to 82.4 weeks)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Topotecan and Bevacizumab: Resistant Participants | Topotecan and Bevacizumab: Sensitive Participants | Topotecan and Bevacizumab: All Participants
Number analyzed (Participants) | 23 | 27 | 50
participants
  CR | 0 | 0 | 0
  PR | 2 | 6 | 8
  SD | 9 | 11 | 20
  PD | 9 | 4 | 13
  Unknown | 3 | 6 | 9

4. Secondary Outcome: Number of Participants With a Tumor Response (CR and PR)
Description: Tumor response was determined using the RECIST guidelines. CR: disappearance of all target lesions. PR: >=30% decrease in sum of LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Baseline to disease progression or death (up to 82.4 weeks)
Population: ITT Population
Measure: Number; unit: participants
Groups:
- Topotecan and Bevacizumab: Sensistive Participants: Participants were to receive oral topotecan 2.3 milligrams (mg)/meters squared (m^2)/day for 5 consecutive days (Days 1 to 5) and intravenous (IV) bevacizumab 15 mg/kilograms (kg) on Day 1 of each 21-day cycle. Treatment was to be continued for up to 8 cycles (a minimum of 4 cycles was recommended) or until disease progression or development of unacceptable toxicity, whichever occurred first. Prior approval from GlaxoSmithKline's study physician was needed for participants who required treatment beyond 8 cycles. The time to progression from the end of prior chemotherapy was >90 days; therefore, these participants were termed "sensitive".
Arm/Group | Topotecan and Bevacizumab: Resistant Participants | Topotecan and Bevacizumab: Sensistive Participants | Topotecan and Bevacizumab: All Participants
Number analyzed (Participants) | 23 | 27 | 50
participants | 2 | 6 | 8

5. Secondary Outcome: Duration of Tumor Response (CR and PR)
Description: Tumor response was determined using the RECIST guidelines. CR: disappearance of all target lesions. PR: >=30% decrease in sum of LD of target lesions, taking as reference the baseline sum LD. Duration of response is defined as the time from start of response (CR or PR) until progression or death due to any cause. For participants who did not progress or die, the time of initiation of post-treatment anti-cancer therapy or the time of last contact was used.
Time Frame: Baseline to disease progression or death (up to 82.4 weeks)
Population: Participants from the ITT Population who had CR and PR
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Topotecan and Bevacizumab
Number analyzed (Participants) | 8
weeks | 20.6 [15.6 to 41.0]

6. Secondary Outcome: Time to Tumor Response (CR and PR)
Description: Tumor response was determined using the RECIST guidelines. CR: disappearance of all target lesions. PR: >=30% decrease in sum of LD of target lesions, taking as reference the baseline sum LD. Time to response is defined as the time from initiation of investigational product to the time of first documented response (CR or PR).
Time Frame: Baseline to disease progression or death (up to 82.4 weeks)
Population: Participants from the ITT Population who had CR and PR
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Topotecan and Bevacizumab
Number analyzed (Participants) | 8
weeks | 5.8 [5.3 to 12.7]

7. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from initiation of investigational product to death due to any cause. For participants who did not die, the time of last contact was used.
Time Frame: Baseline to disease progression or death (up to 82.4 weeks)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Topotecan and Bevacizumab: Resistant Participants | Topotecan and Bevacizumab: Sensitive Participants | Topotecan and Bevacizumab: All Participants
Number analyzed (Participants) | 23 | 27 | 50
weeks | 26.4 [18.1 to 38.0] | 37.0 [30.6 to 48.0] | 32.0 [26.4 to 39.3]

ADVERSE EVENTS:
Groups:
- Topotecan and Bevacizumab: Participants were to receive oral topotecan 2.3 mg/m^2/day for 5 consecutive days (Days 1 to 5) and IV bevacizumab 15 mg/kg on Day 1 of each 21-day cycle. Treatment was to be continued for up to 8 cycles (a minimum of 4 cycles was recommended) or until disease progression or development of unacceptable toxicity, whichever occurred first. Prior approval from GSK's study physician was needed for subjects who required treatment beyond 8 cycles.
Arm/Group | Topotecan and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 18/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topotecan and Bevacizumab (N=50)
Pneumonia (Infections and infestations) | 4
Sepsis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Neutropenic infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 2
Depression (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Topotecan and Bevacizumab (N=50)
Nausea (Gastrointestinal disorders) | 30
Diarrhoea (Gastrointestinal disorders) | 27
Vomiting (Gastrointestinal disorders) | 19
Constipation (Gastrointestinal disorders) | 17
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 4
Oral pain (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 32
Asthenia (General disorders) | 12
Pain (General disorders) | 4
Chills (General disorders) | 3
Gait disturbance (General disorders) | 3
Pyrexia (General disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 27
Neutropenia (Blood and lymphatic system disorders) | 22
Thrombocytopenia (Blood and lymphatic system disorders) | 21
Leukopenia (Blood and lymphatic system disorders) | 11
Pancytopenia (Blood and lymphatic system disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 24
Dehydration (Metabolism and nutrition disorders) | 14
Hypokalaemia (Metabolism and nutrition disorders) | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 6
Hyponatraemia (Metabolism and nutrition disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 10
Headache (Nervous system disorders) | 10
Dysgeusia (Nervous system disorders) | 6
Anxiety (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 6
Confusional state (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 4
Weight decreased (Investigations) | 8
Platelet count decreased (Investigations) | 4
Urinary tract infection (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 6
Proteinuria (Renal and urinary disorders) | 4
Fall (Injury, poisoning and procedural complications) | 3
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.